CLINICAL TRIAL: NCT02497937
Title: A Randomized, Double-blind, Sponsor Un-blinded, Placebo-controlled, Phase 2a Crossover Study to Evaluate the Effect of the TRPV4 Channel Blocker, GSK2798745, on Pulmonary Gas Transfer and Respiration in Patients With Congestive Heart Failure
Brief Title: A Study to Evaluate the Effect of the Transient Receptor Potential Vanilloid 4 (TRPV4) Channel Blocker, GSK2798745, on Pulmonary Gas Transfer and Respiration in Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201881
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
Keywords: GSK2798745; TRPV4 Channel Blocker; Pharmacodynamics; Adults; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — GSK2798745

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2798745 and Placebo (Experimental): Each subject will be randomized to receive GSK2798745 2.4 milligrams (mg) and Placebo once daily for 7 days, each in one of the two treatment periods. Two treatment periods will be separated by a 14-day washout period.
  Interventions: Drug: GSK2798745; Drug: Placebo

INTERVENTIONS:
Drug: GSK2798745 — GSK2798745 will be supplied as granule filled capsule with unit dose strength of 2.4 mg to be administered orally with 240 mL water.
Drug: Placebo — Placebo will be supplied as blend filled capsule to be administered orally with 240 mL water.

SUMMARY:
This study is a single centre, randomised, double-blind, sponsor-unblinded, placebo-controlled, 2 by 2 crossover study in adults with heart failure. In blocking the TRPV4 ion channel and reducing pulmonary interstitial fluid, GSK2798745 may improve pulmonary function, respiration, and gas exchange as well as sleep-disordered breathing in patients with heart failure. Therefore, the current study is designed to investigate the effect of repeat administration of GSK2798745 on pulmonary gas exchange and pulmonary function.

A sufficient number of subjects with heart failure will be enrolled so that 12 subjects complete the two study periods and critical assessments. Subjects will be randomised to receive either GSK2798745 or placebo once daily for a period of 7 days in one treatment period and alternate study medication in the second treatment period. Both the treatment periods will be separated by a washout period of at least 14-days.

This study will consist of a Screening visit within 14 days of the start of Period I and two treatment periods wherein eligible subjects will be randomised to one of the two treatment sequences, a follow-up visit approximately 2 weeks after the completion of second study period. The total duration of the study is approximately 8 weeks from screening to follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* >=21 years of age at the time of signing the informed consent form.
* Diagnosis of heart failure (New York Heart Association Class II-IV) for a minimum of 3 months prior to screening.
* Clinically stable with no changes in optimized guidance-directed medications and no hospitalizations for heart failure for at least 1 month prior to Screening.
* N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) >1000 picogram per milliliter (pg/mL) measured within 6 months prior to OR at Screening.
* Average DLco measurements outside the normal range (percent [%] predicted DLco < 80%) during the Screening Period.
* Body mass index (BMI) >=18 and <=40 kilogram per meter square (kg/m^2).
* Male or female of non-childbearing potential-
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* History of acute coronary syndromes including unstable angina or myocardial infarction within 6 months of screening.
* Coronary revascularization including angioplasty and stenting within 6 months of Screening.
* History of stroke or seizure disorder within 5 years of Screening.
* Diagnosis of asthma.
* Diagnosis of chronic obstructive pulmonary disease (COPD) with FEV1 <50% of predicted measured within 4 weeks of Screening.
* History of a condition that required radiation therapy to the thorax.
* History of any type of malignancy within the past five years with the exception of successfully treated basal cell cancer of the skin.
* Active ulcer disease or gastrointestinal bleeding.
* Current or chronic history of liver disease, known hepatic impairment, or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Alanine transaminase (ALT) >2x Upper Limit of Normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QT interval corrected (QTc) > 450 millisecond (msec) or QTc > 480 msec in subjects with Bundle Branch Block.
* History or current evidence of any serious or clinically significant gastrointestinal, renal, endocrine, neurologic, hematologic or other condition that is uncontrolled on permitted therapies or that would, in the opinion of the investigator or the GlaxoSmithKline (GSK) medical monitor, make the subject unsuitable for inclusion in this study.
* Use of medications specified for the treatment of COPD including short- and long acting bronchodilators (beta-agonists and anticholinergics) and inhaled glucocorticoids as well as oxygen therapy.
* Use of a listed prohibited medication within the restricted timeframe relative to the first dose of study medication.
* Use of a strong inhibitors or inducers of cytochrome P450 (CYP) 3A or p-glycoprotein.
* Current smoker.
* History of drug/substance abuse within the past 2 years.
* History of alcohol abuse within 6 months of the study. Defined as an average weekly alcohol consumption of >14 drinks for men or >7 drinks for women. One drink is equivalent to 12 grams (g) of alcohol: approximately 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine, or 1.5 ounces of (45 mL) 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months of screening. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* Use of another investigational product in a clinical study within the following time period prior to the first administration of study medication in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first administration of study medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, sponsor-unblinded, placebo-controlled, 2 by 2 crossover study in adults with heart failure. A total of 11 participants with Congestive Heart Failure were enrolled in the study. Study was conducted in the United States.
Groups:
- Sequence A (GSK2798745 2.4 mg)/P (Placebo): Eligible participants were randomized to one of two treatment sequences AP and PA where A=GSK2798745 2.4 mg and P=Placebo. In this sequence, participants received GSK2798745 2.4 milligrams (mg) once daily orally with 240 milliliter (mL) water in Period 1 and placebo in Period 2 for 7 days. Treatment periods were separated by a washout period of 14 days.
- Sequence P (Placebo)/A (GSK2798745 2.4 mg): Eligible participants were randomized to one of two treatment sequences AP and PA where A=GSK2798745 2.4 mg and P=Placebo. In this sequence, participants received placebo in Period 1 and GSK2798745 2.4mg once daily orally with 240 mL water in Period 2 for 7 days. Treatment periods were separated by a washout period of 14 days.
Period: Period 1 (Up to 7 Days)
Arm/Group | Sequence A (GSK2798745 2.4 mg)/P (Placebo) | Sequence P (Placebo)/A (GSK2798745 2.4 mg)
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout Period (Up to 14 Days)
Arm/Group | Sequence A (GSK2798745 2.4 mg)/P (Placebo) | Sequence P (Placebo)/A (GSK2798745 2.4 mg)
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Period 2 (Up to 7 Days)
Arm/Group | Sequence A (GSK2798745 2.4 mg)/P (Placebo) | Sequence P (Placebo)/A (GSK2798745 2.4 mg)
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Subjects population comprised of all randomized participants who received at least one dose of study medication.
Groups:
- All Treatment Combined: Eligible participants were randomized to one of two treatment sequences AP and PA where A=GSK2798745 2.4 mg and P=Placebo. In sequence AP, participants received GSK2798745 2.4 milligrams (mg) once daily orally with 240 milliliter (mL) water in Period 1 and placebo in Period 2 for 7 days. In sequence PA, participants received placebo in Period 1 and GSK2798745 2.4mg once daily orally with 240 mL water in Period 2 for 7 days. In both sequence AP and PA, treatment periods were separated by a washout period of 14 days. Data represents all treatments combined.
Arm/Group | All Treatment Combined
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 4
  White | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Diffusing Capacity of the Lung for Carbon Monoxide (DLco) on Pulmonary Gas Transfer (Site: Mayo)
Description: DLco is a measure of the ability of a gas to transfer from alveoli across the alveolar epithelium and capillary endothelium to the red blood cells. Changes in DLco reflect the alveolar-capillary membrane conductance. Acute pulmonary congestion causes a reduction in DLco. In participants with heart failure, decrease in DLco serves as a predictor of disease progression. An impairment in the diffusing capacity of the lung may be related to symptoms and exercise intolerance associated with heart failure. DLco was measured just prior to and after the 3- minute step test on Days -1, and 7 and just prior to and after an intravenous saline infusion on Day 5. Day -1 was Baseline and change from Baseline was calculated from Day -1 pre-exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as Baseline. Data of DLco (milliliter per millimeter of mercury per minute [mL/mmHg/min]) for Mayo site is presented.
Time Frame: Baseline, Day 4, Day 5 and Day 7 of each treatment period
Population: Analysis Population comprised of participants in the 'All Subjects' population having Baseline and post-Baseline assessments of the endpoint of interest for both periods. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: mL/mmHg/min
Groups:
- Placebo: Participants received placebo capsule orally once daily with 240 mL water for a period of 7 days in Periods 1 and 2.
- GSK2798745 2.4 mg: Participants received GSK2798745 2.4 mg capsule orally once daily with 240 mL water for a period of 7 days in Periods 1 and 2.
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 7 | 7
mL/mmHg/min
  Day -1, post exercise,n =7,7 | 0.6 (0.98) | 1.4 (1.47)
  Day 4, n =6,7: number analyzed (Participants) | 6 | 7
  Day 4, n =6,7 | -0.4 (0.85) | 0.6 (1.16)
  Day 5,pre infusion,n =7,7 | -1.0 (0.94) | 0.4 (1.31)
  Day 5,post infusion,n =7,7 | -0.8 (0.65) | -0.7 (0.81)
  Day 7,pre exercise,n =7,7 | -0.6 (1.63) | 0.7 (1.91)
  Day 7,post exercise,n =7,7 | 0.4 (1.38) | 1.6 (2.45)
Statistical Analysis 1: Comparison: Placebo vs GSK2798745 2.4 mg; Test type: Other; Mean Difference (Net) = 0.793, 95% CI 2-sided [-0.925 to 2.512] — Difference estimate of DLco on Day 7 has been presented for Mayo site

2. Primary Outcome: Change From Baseline in the Diffusing Capacity of the Lung for DLco on Pulmonary Gas Transfer (Site: Hennepin)
Description: DLco is a measure of the ability of a gas to transfer from the alveoli across the alveolar epithelium and the capillary endothelium to the red blood cells. Changes in DLco reflect the alveolar-capillary membrane conductance. Acute pulmonary congestion cause a reduction in DLco. In participants with heart failure, decrease in DLco serves as a predictor of disease progression. An impairment in the diffusing capacity of the lung may be related to the symptoms and exercise intolerance associated with heart failure. DLco was measured just prior to and after the 3- minute step test on Days -1, and 7 and just prior to and after an intravenous saline infusion on Day 5. Day -1 was Baseline and change from Baseline was calculated from Day -1 Pre-Exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as the Baseline. Statistical analysis was not performed as the sample size was too small
Time Frame: Baseline, Day 4, Day 5 and Day 7 of each treatment period
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: mL/mmHg/min
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 4 | 4
mL/mmHg/min
  Day -1, post exercise, n =4, 3: number analyzed (Participants) | 4 | 3
  Day -1, post exercise, n =4, 3 | 1.3 (1.32) | 1.0 (0.47)
  Day 4, n =4, 3: number analyzed (Participants) | 4 | 3
  Day 4, n =4, 3 | 1.5 (1.11) | 0.1 (1.05)
  Day 5,pre infusion,n =4,3: number analyzed (Participants) | 4 | 3
  Day 5,pre infusion,n =4,3 | 0.2 (0.53) | -0.3 (0.24)
  Day 5,post infusion,n =4,4 | 0.7 (1.47) | 0.8 (1.31)
  Day 7,pre exercise, n =4,3: number analyzed (Participants) | 4 | 3
  Day 7,pre exercise, n =4,3 | 0.4 (1.82) | -0.6 (1.20)
  Day 7,post exercise, n =4,3: number analyzed (Participants) | 4 | 3
  Day 7,post exercise, n =4,3 | 1.2 (1.01) | 0.4 (1.12)

3. Secondary Outcome: Change From Baseline in Diffusing Capacity of the Lung for Nitric Oxide (DLno) and Membrane Conductance (DM)
Description: DLno is a measure of the ability of a gas to transfer from the alveoli across the alveolar epithelium and the capillary endothelium to the red blood cells. Changes in DLco reflect the alveolar-capillary DM. Since nitric oxide has a greater affinity for hemoglobin, transfer of gas mainly limits the diffusion of nitric oxide across the alveolar capillary membrane. Day -1 was Baseline and change from Baseline was calculated from Day -1 pre-exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as Baseline. The data is presented only for participants from the Mayo Clinic as the data was not collected at Hennepin.
Time Frame: Baseline, Day 4, Day 5 and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/mmHg/min
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 7 | 7
mL/mmHg/min
  DLno,Day -1,post-exercise, n =7, 7 | 2.1 (1.87) | 3.5 (3.66)
  DLno,Day 4, n =6, 7: number analyzed (Participants) | 6 | 7
  DLno,Day 4, n =6, 7 | -2.3 (4.01) | 5.0 (5.51)
  DLno,Day 5,pre-infusion, n =7, 7 | -6.0 (6.50) | 2.4 (8.56)
  DLno,Day 5,post-infusion, n =7, 7 | -2.7 (3.83) | -3.3 (3.27)
  DLno,Day 7,pre-exercise, n =7, 7 | -1.9 (6.19) | 6.0 (9.96)
  DLno,Day 7, post-exercise,n =7,7 | 1.5 (5.37) | 8.6 (10.19)
  DM,Day -1,post-exercise, n =7, 7 | 1.0 (0.85) | 1.7 (1.53)
  DM,Day 4, n =6, 7: number analyzed (Participants) | 6 | 7
  DM,Day 4, n =6, 7 | -1.0 (1.82) | 2.4 (2.61)
  DM,Day 5,pre-infusion, n =7, 7 | -2.7 (2.95) | 1.2 (3.92)
  DM,Day 5,post-infusion, n =7, 7 | -1.2 (1.74) | -1.5 (1.49)
  DM,Day 7,pre-exercise, n =7, 7 | -0.9 (2.81) | 2.8 (4.55)
  DM,Day 7, post-exercise,n =7,7 | 0.7 (2.44) | 4.1 (4.74)

4. Secondary Outcome: Change From Baseline in Capillary Blood Volume (Vc)
Description: Vc is defined as volume of blood within the capillaries. Day -1 was Baseline and change from Baseline was calculated from Day -1 pre-exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as the Baseline. The data is presented only for participants from the Mayo Clinic as the data was not collected at Hennepin.
Time Frame: Baseline, Day 4, Day 5 and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 7 | 7
mL
  Day -1,post exercise, n =7, 7 | 1.6 (8.39) | 10.4 (14.77)
  Day 4, n =6, 7: number analyzed (Participants) | 6 | 7
  Day 4, n =6, 7 | -2.6 (8.64) | -0.2 (9.40)
  Day 5,pre infusion, n =7, 7 | -0.1 (11.60) | 3.0 (12.99)
  Day 5,post infusion, n =7, 7 | -4.9 (14.19) | -2.3 (11.70)
  Day 7,pre exercise, n =7, 7 | -4.7 (12.86) | -2.6 (13.99)
  Day 7, post exercise,n =7,7 | 0.3 (12.33) | 3.3 (15.35)

5. Secondary Outcome: Change From Baseline in DLco Following Exercise and Following an Intravenous Saline Infusion (Site: Mayo)
Description: DLco is a measure of the ability of a gas to transfer from the alveoli across the alveolar epithelium and the capillary endothelium to the red blood cells. Changes in DLco reflect the alveolar-capillary membrane conductance. Acute pulmonary congestion causes a reduction in DLco. In participants with heart failure, decrease in DLco serves as a predictor of disease progression. DLco was measured just prior to and after the 3- minute step test on Days -1, and 7 and just prior to and after an intravenous saline infusion on Day 5. Day -1 was Baseline and change from Baseline was calculated from Day -1 pre-exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as the Baseline. Data for DLco following exercise and following an intravenous saline infusion is presented for Mayo site.
Time Frame: Baseline, Day 5 and Day 7 of each treatment period
Population: Analysis Population.
Measure: Mean (Standard Deviation); unit: mL/mmHg/min
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 7 | 7
mL/mmHg/min
  Day -1,post exercise | 0.6 (0.98) | 1.4 (1.47)
  Day 5,post infusion | -0.8 (0.65) | -0.7 (0.81)
  Day 7, post exercise | 0.4 (1.38) | 1.6 (2.45)

6. Secondary Outcome: Change From Baseline in DLco Following Exercise and Following an Intravenous Saline Infusion (Site: Hennepin)
Description: DLco is a measure of the ability of a gas to transfer from the alveoli across the alveolar epithelium and the capillary endothelium to the red blood cells. Changes in DLco reflect the alveolar-capillary membrane conductance. Acute pulmonary congestion cause a reduction in DLco. In participants with heart failure, decrease in DLco serves as a predictor of disease progression. DLco was measured just prior to and after the 3- minute step test on Days -1, and 7 and just prior to and after an intravenous saline infusion on Day 5. Day -1 was Baseline and change from Baseline was calculated from Day -1 pre-Exercise of the respective period, except when calculating the post-infusion change from Baseline, where the pre-infusion value was used as the Baseline. Data for DLco following exercise and following an intravenous saline infusion is presented for Hennepin site is presented.
Time Frame: Baseline, Day 5 and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/mmHg/min
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 4 | 4
mL/mmHg/min
  Day -1,post exercise,n=4,3: number analyzed (Participants) | 4 | 3
  Day -1,post exercise,n=4,3 | 1.3 (1.32) | 1.0 (0.47)
  Day 5,post infusion,n=4,4 | 0.7 (1.47) | 0.8 (1.31)
  Day 7, post exercise,n=4,3: number analyzed (Participants) | 4 | 3
  Day 7, post exercise,n=4,3 | 1.2 (1.01) | 0.4 (1.12)

7. Secondary Outcome: Change From Baseline in the Ventilation/Volume of Carbon Dioxide Production (VE/VCO2) Ratio
Description: Participants were asked to participate in a submaximal exercise test that consisted of 3 parts: a 2-minute (min) resting Baseline, a 3-min step exercise and a 1-min recovery period. Throughout the test, breathing pattern, gas exchange, and heart rate were monitored using a simplified gas analysis system. Respiratory exchange ratio and the Borg Rating of Perceived Exertion measures were utilized to ensure participants perform progressive exercise while maintaining a submaximal level throughout the exercise period. Minute ventilation, breath frequency, tidal volume, oxygen consumption, carbon dioxide (CO2) production, Respiratory exchange ratio (RER) and end tidal CO2 were obtained from the breath-by-breath gas measurements. The VE/VCO2 slope and other variables were derived from this data. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and Day 7 of each treatment period
Population: Analysis Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Ratio
  Period 1 Day -1,post 1 min | 1.3 (3.1) | 0.3 (5.0)
  Period 1 Day -1,at rest,post 2 min | 1.6 (6.40) | 1.8 (11.93)
  Period 1 Day -1,post 3 min | 0.7 (9.15) | -4.5 (6.68)
  Period 1 Day -1,recovery | -5.1 (4.17) | -5.7 (4.31)
  Period 1 Day 7,at rest | 2.4 (10.1) | 0.6 (2.1)
  Period 1 Day 7,post 1 min | 0.7 (10.1) | 0.0 (3.8)
  Period 1 Day 7,post 2 min | -1.2 (11.99) | 1.6 (10.37)
  Period 1 Day 7,post 3 min | 1.6 (13.29) | -1.2 (3.97)
  Period 1 Day 7,recovery | -8.0 (5.68) | -5.4 (3.26)
  Period 2 Day -1,post 1 min | -3.6 (4.1) | -2.1 (4.5)
  Period 2 Day -1,post 2 min | -3.7 (4.68) | -2.8 (5.74)
  Period 2 Day -1,post 3 min | -4.7 (6.65) | -4.2 (5.86)
  Period 2 Day -1,Recovery | -9.3 (3.04) | -7.6 (6.13)
  Period 2 Day 7 at rest | -2.5 (6.3) | -0.9 (4.2)
  Period 2 Day 7,post 1 min | -4.0 (4.4) | -2.5 (3.7)
  Period 2 Day 7,post 2 min | -2.6 (4.16) | -3.9 (4.98)
  Period 2 Day 7,post 3 min | -0.7 (10.21) | -6.4 (3.65)
  Period 2 Day 7,Recovery | -2.1 (22.58) | -7.6 (5.17)

8. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 Second (FEV1), Forced Expiratory Flows (FEF) 25-75, FEF50 and FEF75
Description: FEV1 was defined as the volume of air that can be forced out in one second after taking a deep breath. FVC is the total amount of air exhaled during the lung function test. FEF is the the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. FEF 25-75, FEF50 and FEF75 is defined as a reduction in forced expiratory flow at 25 to 75 percent of the pulmonary volume. Results presented combines data across all sites. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline, Day 4 and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Liters
  FVC,Day 4,n=10,11: number analyzed (Participants) | 10 | 11
  FVC,Day 4,n=10,11 | -0.0 (0.11) | -0.1 (0.10)
  FVC,Day 7,n=11,11 | -0.0 (0.10) | -0.0 (0.19)
  FEV1,Day 4,n=10,11: number analyzed (Participants) | 10 | 11
  FEV1,Day 4,n=10,11 | -0.1 (0.09) | -0.0 (0.09)
  FEV1,Day 7,n=11,11 | -0.1 (0.08) | -0.0 (0.12)
  FEF 25-75,Day 4,n=10,11: number analyzed (Participants) | 10 | 11
  FEF 25-75,Day 4,n=10,11 | -0.2 (0.26) | 0.1 (0.34)
  FEF 25-75,Day 7,n=11,11 | -0.1 (0.16) | -0.1 (0.25)
  FEF50,Day 4,n=10,11: number analyzed (Participants) | 10 | 11
  FEF50,Day 4,n=10,11 | -0.3 (0.36) | 0.0 (0.43)
  FEF50,Day 7,n=11,11 | -0.2 (0.30) | -0.0 (0.32)
  FEF75,Day 4,n=10,11: number analyzed (Participants) | 10 | 11
  FEF75,Day 4,n=10,11 | -0.0 (0.08) | 0.0 (0.14)
  FEF75,Day 7,n=11,11 | -0.0 (0.06) | -0.0 (0.10)

9. Secondary Outcome: Change From Baseline in Functional Residual Capacity (FRC)
Description: FRC is the volume of air present in the lungs at the end of passive expiration. FRC was planned to be measured by body plethysmography. Analysis was planned but not performed. FRC parameter was not collected because other measures which were collected served as reasonable surrogates.
Time Frame: Baseline, Day 4 and Day 7 of each treatment period
Population: Analysis Population. Analysis was planned but not performed. FRC parameter was not collected because other measures which were collected served as reasonable surrogates.
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in End-expiratory Lung Volume (EELV) Measured by Body Plethysmograph
Description: EELV corresponds to FRC in the presence of positive end expiration pressure (PEEP). Analysis was planned but not performed. EELV parameter was not collected because other measures which were collected served as reasonable surrogates.
Time Frame: Baseline, Day 4 and Day 7 of each treatment period
Population: Analysis Population. Analysis was planned but not performed. EELV parameter was not collected because other measures which were collected served as reasonable surrogates.
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Dyspnea Score
Description: Dyspnea was assessed using a standardized, validated 5-point Likert scale. Participants were asked to check the box next to the statement that most accurately described their current state of breathlessness or shortness of breath. Scale consisted of 5 points : 1- Not short of breath, 2- Mildly short of breath, 3- Moderately short of breath, 4- Severely short of breath and 5- Very severely short of breath. Participants rated their current state of breathlessness on this 5 point scale. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point .
Time Frame: Baseline, Day 5 and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Scores on a scale
  Period 1 Day-1,post exercise,n=4,2: number analyzed (Participants) | 4 | 2
  Period 1 Day-1,post exercise,n=4,2 | 0.5 (0.58) | 0.5 (0.71)
  Period 1 Day5,pre infusion,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1 Day5,pre infusion,n=5,6 | 0.2 (0.45) | -0.2 (0.41)
  Period 1 Day5,pre infusion-Orthopnea,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1 Day5,pre infusion-Orthopnea,n=5,6 | 0.2 (0.45) | -0.2 (0.41)
  Period 1 Day7,pre exercise,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1 Day7,pre exercise,n=5,6 | 0.0 (0.00) | 0.0 (0.63)
  Period 1 Day7,post exercise,n=3,2: number analyzed (Participants) | 3 | 2
  Period 1 Day7,post exercise,n=3,2 | 1.3 (2.31) | 0.5 (0.71)
  Period 2 Day -1,post exercise,n=2,3: number analyzed (Participants) | 2 | 3
  Period 2 Day -1,post exercise,n=2,3 | 2.0 (2.83) | 1.3 (1.15)
  Period 2 Day5,pre infusion,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2 Day5,pre infusion,n=6,5 | -0.3 (1.03) | -0.2 (1.10)
  Period 2 Day5,pre infusion-Orthopnea,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2 Day5,pre infusion-Orthopnea,n=6,5 | -0.3 (1.03) | -0.4 (0.89)
  Period 2 Day7,pre exercise,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2 Day7,pre exercise,n=6,5 | -0.5 (0.84) | -0.4 (0.89)
  Period 2 Day7,post exercise,n=3,4: number analyzed (Participants) | 3 | 4
  Period 2 Day7,post exercise,n=3,4 | -1.0 (1.00) | 0.3 (1.71)

12. Secondary Outcome: Respiratory Rate Over Time Continuously Measured by Body Sensor (Site: Mayo Only)
Description: Continuous remote monitoring was performed during each 7-day study period utilizing the Preventice BodyGuardian Remote Monitoring System. Participants were instructed to wear the sensor throughout each study period. Respiratory monitoring data was collected in different body positions like standing, leaning, lying and unknown. Data is presented only for participants from Mayo clinic.
Time Frame: Up to Day 7 of each treatment period
Population: All Subjects population comprised of all randomized participants who received at least one dose of study medication. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 7 | 7
breaths per minute
  Day -1,Not set,n=4,3: number analyzed (Participants) | 4 | 3
  Day -1,Not set,n=4,3 | 22.9 (5.14) | 13.3 (1.58)
  Day -1,Standing,n=4,4: number analyzed (Participants) | 4 | 4
  Day -1,Standing,n=4,4 | 15.3 (2.79) | 16.8 (3.43)
  Day -1,Leaning,n=5,4: number analyzed (Participants) | 5 | 4
  Day -1,Leaning,n=5,4 | 15.4 (3.06) | 17.7 (3.56)
  Day -1,Lying,n=4,4: number analyzed (Participants) | 4 | 4
  Day -1,Lying,n=4,4 | 17 (3.08) | 15.6 (2.26)
  Day -1,Unknown,n=0,2: number analyzed (Participants) | 0 | 2
  Day -1,Unknown,n=0,2 |  | 17.5 (3.75)
  Day 4,Not set,n=6,3: number analyzed (Participants) | 6 | 3
  Day 4,Not set,n=6,3 | 14.9 (3.64) | 13.8 (1.09)
  Day 4,Standing,n=6,6: number analyzed (Participants) | 6 | 6
  Day 4,Standing,n=6,6 | 15.9 (3.39) | 15.5 (3.1)
  Day 4,Leaning,n=6,6: number analyzed (Participants) | 6 | 6
  Day 4,Leaning,n=6,6 | 18.6 (4.19) | 17.9 (3.94)
  Day 4,Lying,n=6,5: number analyzed (Participants) | 6 | 5
  Day 4,Lying,n=6,5 | 16.8 (3.6) | 16.5 (3.41)
  Day 4,Unknown,n=2,3: number analyzed (Participants) | 2 | 3
  Day 4,Unknown,n=2,3 | 15.5 (2.18) | 13.2 (3.54)
  Day 7,Not set,n=3,4: number analyzed (Participants) | 3 | 4
  Day 7,Not set,n=3,4 | 15.7 (3.88) | 15.1 (2.76)
  Day 7,Standing,n=7,4: number analyzed (Participants) | 7 | 4
  Day 7,Standing,n=7,4 | 15.9 (3.54) | 15.5 (3.53)
  Day 7,Leaning,n=6,4: number analyzed (Participants) | 6 | 4
  Day 7,Leaning,n=6,4 | 15.7 (3.89) | 17.5 (3.68)
  Day 7,Lying,n=7,4: number analyzed (Participants) | 7 | 4
  Day 7,Lying,n=7,4 | 16.8 (3.88) | 16 (3.6)

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure(SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in a semi-supine position after 5 minutes rest at Baseline and up to 7 days of each treatment period. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: All Subjects Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Millimeters of mercury
  SBP,Period 1, Day 1,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 1,n=5,6 | -6.8 (7.12) | 2.5 (19.56)
  SBP,Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 2,n=5,6 | -7.8 (13.86) | -2.5 (12.49)
  SBP,Period 1, Day 3,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 3,n=5,6 | -8.8 (12.52) | 0.0 (10.41)
  SBP,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 4,n=5,6 | -9.2 (9.71) | 0.8 (14.66)
  SBP,Period 1, Day 5,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 5,n=5,6 | -10.4 (11.78) | 0.3 (24.91)
  SBP,Period 1, Day 6,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 6,n=5,6 | -12.8 (7.05) | 0.0 (14.85)
  SBP,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  SBP,Period 1, Day 7,n=5,6 | -3.2 (18.74) | 9.0 (25.17)
  SBP,Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 1,n=6,5 | -14.0 (22.45) | -9.2 (17.33)
  SBP,Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 2,n=6,5 | -12.7 (31.65) | -6.4 (15.92)
  SBP,Period 2, Day 3,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 3,n=6,5 | -14.5 (34.88) | -8.0 (11.75)
  SBP,Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 4,n=6,5 | -13.5 (25.62) | -4.4 (14.05)
  SBP,Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 5,n=6,5 | -19.0 (23.10) | -10.8 (14.57)
  SBP,Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 6,n=6,5 | -12.5 (16.38) | -7.4 (10.57)
  SBP,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  SBP,Period 2, Day 7,n=6,5 | -11.5 (27.57) | -2.2 (14.36)
  DBP,Period 1, Day 1,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 1,n=5,6 | -3.4 (10.14) | 0.3 (12.06)
  DBP,Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 2,n=5,6 | -7.6 (8.02) | -4.0 (14.03)
  DBP,Period 1, Day 3,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 3,n=5,6 | -14.6 (4.83) | -0.3 (9.99)
  DBP,Period 1,Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1,Day 4,n=5,6 | -5.0 (9.62) | -4.3 (12.21)
  DBP,Period 1, Day 5,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 5,n=5,6 | -8.0 (8.03) | -5.8 (11.20)
  DBP,Period 1, Day 6,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 6,n=5,6 | -9.8 (5.67) | 0.2 (8.23)
  DBP,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  DBP,Period 1, Day 7,n=5,6 | 0.2 (13.01) | 6.5 (12.00)
  DBP,Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 1,n=6,5 | -9.2 (13.91) | 0.4 (9.50)
  DBP,Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 2,n=6,5 | -9.7 (18.41) | -8.0 (8.43)
  DBP,Period 2, Day 3,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 3,n=6,5 | -7.2 (20.47) | -2.0 (6.82)
  DBP,Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 4,n=6,5 | -9.8 (12.27) | 1.2 (12.79)
  DBP,Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 5,n=6,5 | -10.7 (15.38) | -3.6 (8.41)
  DBP,Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 6,n=6,5 | -8.2 (11.62) | 5.2 (9.26)
  DBP,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  DBP,Period 2, Day 7,n=6,5 | -9.3 (13.95) | 1.2 (11.03)

14. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a semi-supine position after 5 minutes rest at Baseline and up to 7 days of each treatment period. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
beats per minute
  Period 1, Day 1,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 1,n=5,6 | -7.0 (7.42) | 5.2 (11.46)
  Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 2,n=5,6 | -5.8 (5.36) | -2.8 (15.72)
  Period 1, Day 3,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 3,n=5,6 | -2.4 (9.21) | -0.8 (17.60)
  Period 1,Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1,Day 4,n=5,6 | -4.6 (10.16) | -4.0 (16.84)
  Period 1, Day 5,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 5,n=5,6 | -4.8 (7.79) | 2.2 (6.31)
  Period 1, Day 6,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 6,n=5,6 | -6.2 (5.81) | 0.8 (4.12)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | -3.2 (7.95) | 5.2 (5.08)
  Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 1,n=6,5 | -7.3 (9.46) | 7.0 (9.08)
  Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 2,n=6,5 | -8.0 (15.80) | -1.0 (2.35)
  Period 2, Day 3,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 3,n=6,5 | -7.5 (16.34) | -4.0 (4.80)
  Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4,n=6,5 | -9.0 (13.52) | 0.6 (5.86)
  Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 5,n=6,5 | -11.0 (15.67) | 0.2 (4.15)
  Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 6,n=6,5 | -11.0 (16.46) | 2.2 (9.04)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | -11.2 (14.46) | -1.2 (10.52)

15. Secondary Outcome: Change From Baseline in Respiration Rate
Description: Respiration rate was measured in a semi-supine position after 5 minutes rest at Baseline and up to 7 days of each treatment period. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
breaths per minute
  Period 1, Day 1,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 1,n=5,6 | 0.6 (0.89) | 1.0 (3.95)
  Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 2,n=5,6 | -0.2 (2.86) | 0.7 (3.01)
  Period 1, Day 3,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 3,n=5,6 | 0.2 (1.79) | 2.0 (3.46)
  Period 1,Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1,Day 4,n=5,6 | 0.6 (1.67) | 0.8 (1.79)
  Period 1, Day 5,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 5,n=5,6 | 1.2 (2.59) | 1.8 (4.58)
  Period 1, Day 6,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 6,n=5,6 | -0.2 (3.63) | 2.0 (3.10)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | 1.2 (4.38) | 1.7 (3.44)
  Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 1,n=6,5 | 2.3 (3.67) | 1.0 (3.74)
  Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 2,n=6,5 | 2.7 (2.73) | 3.2 (2.39)
  Period 2, Day 3,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 3,n=6,5 | 1.7 (3.88) | 3.0 (2.00)
  Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4,n=6,5 | 1.7 (3.67) | 4.6 (3.58)
  Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 5,n=6,5 | 2.3 (3.44) | 1.0 (3.00)
  Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 6,n=6,5 | 2.7 (1.03) | 2.6 (2.41)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | 1.0 (2.45) | -1.0 (1.73)

16. Secondary Outcome: Change From Baseline in Temperature
Description: Body temperature was measured in a semi-supine position after 5 minutes rest at Baseline and up to 7 days of each treatment period. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Celsius
  Period 1, Day 1,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 1,n=5,6 | -0.2 (0.55) | -0.0 (0.10)
  Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 2,n=5,6 | -0.1 (0.16) | -0.0 (0.24)
  Period 1, Day 3,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 3,n=5,6 | 0.0 (0.15) | -0.0 (0.33)
  Period 1,Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1,Day 4,n=5,6 | 0.2 (0.34) | -0.2 (0.12)
  Period 1, Day 5,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 5,n=5,6 | -0.1 (0.11) | -0.1 (0.19)
  Period 1, Day 6,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 6,n=5,6 | 0.0 (0.30) | -0.1 (0.32)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | -0.0 (0.16) | -0.2 (0.29)
  Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 1,n=6,5 | 0.2 (0.55) | 0.1 (0.13)
  Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 2,n=6,5 | 0.2 (0.44) | -0.0 (0.28)
  Period 2, Day 3,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 3,n=6,5 | 0.0 (0.49) | -0.1 (0.21)
  Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4,n=6,5 | 0.1 (0.46) | -0.2 (0.21)
  Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 5,n=6,5 | -0.2 (0.26) | -0.1 (0.19)
  Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 6,n=6,5 | 0.1 (0.42) | -0.1 (0.24)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | 0.1 (0.39) | 0.1 (0.21)

17. Secondary Outcome: Change From Baseline in Percent Oxygen in Blood
Description: Percent oxygen in blood was measured using pulse oximetry in a semi-supine position after 5 minutes rest at Baseline and up to 7 days of each treatment period. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage of oxygen
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Percentage of oxygen
  Period 1, Day 1,n=4,6: number analyzed (Participants) | 4 | 6
  Period 1, Day 1,n=4,6 | 0.0 (0.82) | -0.3 (1.37)
  Period 1, Day 2,n=4,5: number analyzed (Participants) | 4 | 5
  Period 1, Day 2,n=4,5 | 1.3 (0.96) | -1.2 (0.84)
  Period 1, Day 3,n=3,6: number analyzed (Participants) | 3 | 6
  Period 1, Day 3,n=3,6 | 0.7 (1.53) | -0.7 (1.75)
  Period 1,Day 4,n=4,6: number analyzed (Participants) | 4 | 6
  Period 1,Day 4,n=4,6 | 0.3 (0.96) | 0.0 (1.10)
  Period 1, Day 5,n=4,6: number analyzed (Participants) | 4 | 6
  Period 1, Day 5,n=4,6 | 1.0 (1.63) | 0.5 (2.66)
  Period 1, Day 6,n=4,6: number analyzed (Participants) | 4 | 6
  Period 1, Day 6,n=4,6 | 0.3 (0.96) | -0.2 (1.72)
  Period 1, Day 7,n=4,6: number analyzed (Participants) | 4 | 6
  Period 1, Day 7,n=4,6 | -0.3 (1.71) | -0.3 (1.51)
  Period 2, Day 1,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 1,n=6,5 | -1.0 (2.83) | -0.6 (1.82)
  Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 2,n=6,5 | 0.2 (2.99) | 0.0 (1.22)
  Period 2, Day 3,n=6,4: number analyzed (Participants) | 6 | 4
  Period 2, Day 3,n=6,4 | -0.8 (2.64) | -0.3 (2.36)
  Period 2, Day 4,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4,n=6,5 | -1.0 (2.61) | 1.4 (1.82)
  Period 2, Day 5,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 5,n=6,5 | -0.2 (1.33) | 0.2 (1.30)
  Period 2, Day 6,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 6,n=6,5 | -0.5 (2.17) | 0.2 (1.79)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | 0.2 (2.04) | 0.0 (1.87)

18. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECG was obtained using an automated ECG machine at Baseline (Day-1) and single ECG measurements (M) were taken on Day 4 and Day 7. Data for number of participants with abnormal-clinically significant (CS) and abnormal-not clinically significant (NCS) ECG data is presented.
Time Frame: Up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Participants
  Period 1, Day -1, M1, NCS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M1, NCS,n=5,6 | 5 | 6
  Period 1, Day -1, M1, CS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M1, CS,n=5,6 | 0 | 0
  Period 1, Day -1, M2, NCS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M2, NCS,n=5,6 | 5 | 6
  Period 1, Day -1, M2, CS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M2, CS,n=5,6 | 0 | 0
  Period 1, Day -1, M3, NCS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M3, NCS,n=5,6 | 5 | 6
  Period 1, Day -1, M3, CS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day -1, M3, CS,n=5,6 | 0 | 0
  Period 1, Day 4, NCS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 4, NCS,n=5,6 | 5 | 6
  Period 1, Day 4, CS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 4, CS,n=5,6 | 0 | 0
  Period 1, Day 7, NCS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7, NCS,n=5,6 | 5 | 6
  Period 1, Day 7, CS,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7, CS,n=5,6 | 0 | 0
  Period 2, Day -1, M1, NCS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day -1, M1, NCS,n=6,5 | 6 | 5
  Period 2 Day -1, M1, CS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2 Day -1, M1, CS,n=6,5 | 0 | 0
  Period 2, Day -1, M2, NCS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day -1, M2, NCS,n=6,5 | 6 | 5
  Period 2, Day -1, M2, CS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day -1, M2, CS,n=6,5 | 0 | 0
  Period 2, Day -1, M3, NCS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day -1, M3, NCS,n=6,5 | 6 | 5
  Period 2, Day -1, M3, CS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day -1, M3, CS,n=6,5 | 0 | 0
  Period 2, Day 4, NCS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4, NCS,n=6,5 | 6 | 5
  Period 2, Day 4, CS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 4, CS,n=6,5 | 0 | 0
  Period 2, Day 7, NCS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7, NCS,n=6,5 | 6 | 5
  Period 2, Day 7, CS,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7, CS,n=6,5 | 0 | 0

19. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase, Gamma Glutamyl Transferase (GGT) Values
Description: Blood samples were collected to analyze the chemistry parameters including ALT, ALP, AST, creatine kinase and GGT. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
International units per liter
  ALT,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  ALT,Period 1, Day 4,n=5,6 | -1.8 (1.92) | -5.5 (10.41)
  ALT,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  ALT,Period 1, Day 7,n=5,6 | -1.2 (2.77) | -6.2 (8.80)
  ALT,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  ALT,Period 2, Day 4,n=5,5 | 2.8 (5.59) | -3.6 (2.88)
  ALT,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  ALT,Period 2, Day 7,n=6,5 | 5.3 (6.50) | -2.6 (2.70)
  ALP,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  ALP,Period 1, Day 4,n=5,6 | 0.6 (6.54) | -17.8 (35.65)
  ALP,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  ALP,Period 1, Day 7,n=5,6 | -1.0 (7.00) | -15.2 (30.96)
  ALP,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  ALP,Period 2, Day 4,n=5,5 | 0.4 (6.73) | -0.8 (2.39)
  ALP,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  ALP,Period 2, Day 7,n=6,5 | 8.0 (21.46) | 1.2 (6.30)
  AST,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  AST,Period 1, Day 4,n=5,6 | -4.0 (4.80) | -6.7 (9.65)
  AST,Period 1, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  AST,Period 1, Day 7,n=5,5 | -3.2 (3.56) | -7.2 (8.04)
  AST,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  AST,Period 2, Day 4,n=5,5 | 0.0 (9.97) | -8.0 (2.92)
  AST,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  AST,Period 2, Day 7,n=6,5 | 4.2 (7.00) | -4.8 (1.92)
  GGT,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  GGT,Period 1, Day 4,n=5,6 | -6.0 (6.86) | -12.5 (20.71)
  GGT,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  GGT,Period 1, Day 7,n=5,6 | -9.8 (11.82) | -9.5 (11.06)
  GGT,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  GGT,Period 2, Day 4,n=5,5 | 5.8 (16.95) | -4.8 (7.73)
  GGT,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  GGT,Period 2, Day 7,n=6,5 | 9.0 (22.09) | -5.2 (5.54)
  Creatine kinase,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Creatine kinase,Period 1, Day 4,n=5,6 | -57.4 (90.68) | -27.7 (36.14)
  Creatine kinase,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Creatine kinase,Period 1, Day 7,n=5,6 | -64.0 (105.02) | -19.5 (54.42)
  Creatine kinase,Period 2, Day 4,n=5,4: number analyzed (Participants) | 5 | 4
  Creatine kinase,Period 2, Day 4,n=5,4 | -18.0 (25.03) | -59.0 (68.33)
  Creatine kinase,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Creatine kinase,Period 2, Day 7,n=6,5 | -15.8 (22.05) | -47.8 (29.20)

20. Secondary Outcome: Change From Baseline in Albumin and Total Protein Values
Description: Blood samples were collected to analyze the chemistry parameters including albumin and total protein. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Grams per liter
  Albumin,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Albumin,Period 1, Day 4,n=5,6 | -1.6 (1.52) | -0.5 (2.59)
  Albumin,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Albumin,Period 1, Day 7,n=5,6 | -0.6 (2.30) | -0.3 (1.75)
  Albumin,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Albumin,Period 2, Day 4,n=5,5 | -0.4 (0.55) | -0.2 (1.79)
  Albumin,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Albumin,Period 2, Day 7,n=6,5 | 0.2 (1.83) | 0.8 (1.30)
  Total protein,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Total protein,Period 1, Day 4,n=5,6 | -1.0 (5.15) | -1.5 (5.36)
  Total protein,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Total protein,Period 1, Day 7,n=5,6 | 0.8 (5.22) | -1.2 (4.17)
  Total protein,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Total protein,Period 2, Day 4,n=5,5 | -1.6 (2.07) | 0.4 (3.58)
  Total protein,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Total protein,Period 2, Day 7,n=6,5 | -0.8 (3.54) | 2.8 (1.64)

21. Secondary Outcome: Change From Baseline in Chemistry: Calcium, Chloride, Glucose, Potassium, Sodium, Urea/Blood Urea Nitrogen (BUN)
Description: Blood samples were collected to analyze the chemistry parameters including Calcium, Chloride, Glucose, Potassium, Sodium, Urea/BUN. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Millimoles per liter
  Calcium,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Calcium,Period 1, Day 4,n=5,6 | 0.01497 (0.080074) | -0.06653 (0.187817)
  Calcium,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Calcium,Period 1, Day 7,n=5,6 | 0.05988 (0.120434) | -0.05822 (0.185817)
  Calcium,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Calcium,Period 2, Day 4,n=5,5 | -0.05489 (0.020875) | 0.00998 (0.041749)
  Calcium,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Calcium,Period 2, Day 7,n=6,5 | -0.06238 (0.071880) | 0.02994 (0.044632)
  Chloride,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Chloride,Period 1, Day 4,n=5,6 | -1.8 (1.48) | -1.3 (1.97)
  Chloride,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Chloride,Period 1, Day 7,n=5,6 | -1.0 (1.87) | 0.5 (1.76)
  Chloride,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Chloride,Period 2, Day 4,n=5,5 | -0.8 (1.79) | -2.0 (2.35)
  Chloride,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Chloride,Period 2, Day 7,n=6,5 | -2.0 (4.82) | -2.4 (1.82)
  Glucose,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Glucose,Period 1, Day 4,n=5,6 | 3.63035 (4.132346) | 2.04462 (3.557566)
  Glucose,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Glucose,Period 1, Day 7,n=5,6 | 2.04277 (2.486018) | 0.61986 (5.924289)
  Glucose,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Glucose,Period 2, Day 4,n=5,5 | 1.68750 (2.144009) | 3.96341 (3.372569)
  Glucose,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Glucose,Period 2, Day 7,n=6,5 | 1.51727 (4.849639) | 1.23232 (2.196471)
  Potassium,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Potassium,Period 1, Day 4,n=5,6 | 0.22 (0.319) | 0.33 (0.388)
  Potassium,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Potassium,Period 1, Day 7,n=5,6 | 0.16 (0.270) | 0.35 (0.619)
  Potassium,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Potassium,Period 2, Day 4,n=5,5 | 0.04 (0.397) | 0.26 (0.270)
  Potassium,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Potassium,Period 2, Day 7,n=6,5 | -0.23 (0.592) | 0.14 (0.378)
  Sodium,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Sodium,Period 1, Day 4,n=5,6 | -1.0 (4.00) | -2.0 (1.55)
  Sodium,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Sodium,Period 1, Day 7,n=5,6 | -1.4 (3.36) | -1.2 (2.48)
  Sodium,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Sodium,Period 2, Day 4,n=5,5 | -1.0 (1.58) | -0.8 (2.59)
  Sodium,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Sodium,Period 2, Day 7,n=6,5 | -2.2 (2.32) | -1.6 (1.67)
  Urea/BUN,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Urea/BUN,Period 1, Day 4,n=5,6 | -0.0714 (1.34528) | 2.2610 (3.82285)
  Urea/BUN,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Urea/BUN,Period 1, Day 7,n=5,6 | -0.4284 (1.86188) | -0.1785 (2.17448)
  Urea/BUN,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Urea/BUN,Period 2, Day 4,n=5,5 | -1.2852 (3.02504) | -0.5712 (2.53193)
  Urea/BUN,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Urea/BUN,Period 2, Day 7,n=6,5 | -0.2975 (4.41537) | 0.0714 (2.84930)

22. Secondary Outcome: Change From Baseline in Creatinine, Direct Bilirubin, Total Bilirubin, Uric Acid
Description: Blood samples were collected to analyze the chemistry parameters including Creatinine, Direct Bilirubin, Total Bilirubin and Uric acid. Change from Baseline was presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 of each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Micromoles per liter
  Creatinine,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Creatinine,Period 1, Day 4,n=5,6 | -8.1328 (17.06601) | 11.4920 (29.13179)
  Creatinine,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Creatinine,Period 1, Day 7,n=5,6 | -13.2600 (15.91200) | -9.4293 (12.58472)
  Creatinine,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Creatinine,Period 2, Day 4,n=5,5 | -6.0112 (12.84693) | -2.6520 (14.83172)
  Creatinine,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Creatinine,Period 2, Day 7,n=6,5 | -4.8620 (26.95113) | 3.7128 (11.43064)
  Direct Bilirubin,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Direct Bilirubin,Period 1, Day 4,n=5,6 | -0.684 (0.9366) | -0.572 (0.8856)
  Direct Bilirubin,Period 1, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Direct Bilirubin,Period 1, Day 7,n=5,5 | -0.342 (0.7647) | -0.344 (1.4331)
  Direct Bilirubin,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Direct Bilirubin,Period 2, Day 4,n=5,5 | -0.340 (0.7659) | -1.026 (1.5295)
  Direct Bilirubin,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Direct Bilirubin,Period 2, Day 7,n=6,5 | -0.285 (0.6981) | -0.684 (0.9366)
  Total Bilirubin,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Total Bilirubin,Period 1, Day 4,n=5,6 | 1.368 (2.8098) | -1.425 (1.6813)
  Total Bilirubin,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Total Bilirubin,Period 1, Day 7,n=5,6 | 0.684 (1.9497) | 0.002 (2.1646)
  Total Bilirubin,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Total Bilirubin,Period 2, Day 4,n=5,5 | -0.000 (3.1991) | -5.472 (9.2403)
  Total Bilirubin,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Total Bilirubin,Period 2, Day 7,n=6,5 | -0.285 (1.9991) | -5.130 (10.1885)
  Uric acid,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Uric acid,Period 1, Day 4,n=5,6 | -17.8440 (35.43930) | 18.8353 (47.19830)
  Uric acid,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Uric acid,Period 1, Day 7,n=5,6 | -42.8256 (40.20954) | -29.7400 (51.57983)
  Uric acid,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Uric acid,Period 2, Day 4,n=5,5 | -17.8440 (29.44110) | -1.1896 (24.66807)
  Uric acid,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Uric acid,Period 2, Day 7,n=6,5 | 25.7747 (111.31927) | 9.5168 (19.99448)

23. Secondary Outcome: Change From Baseline in Digoxin Level
Description: Blood samples were collected to analyze the digoxin levels. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the baseline value from specified time point value. NA indicates data not available. Standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Nanomoles per liter
  Period 1 Day 1,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 1,n=3,1 | -0.17080 (0.322378) | 0.38430 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 2,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 2,n=3,1 | 0.17080 (0.073959) | 0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 3,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 3,n=3,1 | 0.12810 (0.128100) | 0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 4,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 4,n=3,1 | -0.10248 (0.419417) | 0.12810 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 5,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 5,n=3,1 | 0.25620 (0.221876) | 0.38430 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 6,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 6,n=3,1 | 0.17080 (0.147917) | 0.00000 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1 Day 7,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1 Day 7,n=3,1 | -0.00000 (0.128100) | 0.00000 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 2 Day 1,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 1,n=1,3 | -0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.34160 (0.266661)
  Period 2 Day 2,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 2,n=1,3 | -0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.46970 (0.295834)
  Period 2 Day 3,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 3,n=1,3 | -0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.17080 (0.195676)
  Period 2 Day 4,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 4,n=1,3 | -0.38430 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.42700 (0.195676)
  Period 2 Day 5,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 5,n=1,3 | -0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.25620 (0.128100)
  Period 2 Day 6,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 6,n=1,3 | -0.12810 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.29890 (0.391352)
  Period 2 Day 7,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2 Day 7,n=1,3 | -0.25620 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.42700 (0.369793)

24. Secondary Outcome: Change From Baseline in Troponin I Levels and Type I Collagen Cross-linked C-telopeptide
Description: Blood samples were collected to analyze the troponin I level and type I collagen cross-linked C-telopeptide (T1CCT). Change from Baseline was presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from value at specified time point.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Microgram per liter
  Troponin I,Period 1, Day 2,n=5,6: number analyzed (Participants) | 5 | 6
  Troponin I,Period 1, Day 2,n=5,6 | -0.0044 (0.00658) | -0.0007 (0.00516)
  Troponin I,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Troponin I,Period 1, Day 4,n=5,6 | -0.0118 (0.01117) | -0.0008 (0.00492)
  Troponin I,Period 1, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Troponin I,Period 1, Day 7,n=5,5 | -0.0112 (0.01314) | -0.0056 (0.00876)
  Troponin I,Period 2, Day 2,n=6,5: number analyzed (Participants) | 6 | 5
  Troponin I,Period 2, Day 2,n=6,5 | 0.0023 (0.00898) | 0.0002 (0.00672)
  Troponin I,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Troponin I,Period 2, Day 4,n=5,5 | -0.0036 (0.00498) | -0.0000 (0.01225)
  Troponin I,Period 2, Day 7,n=6,4: number analyzed (Participants) | 6 | 4
  Troponin I,Period 2, Day 7,n=6,4 | -0.0012 (0.01132) | 0.0043 (0.01902)
  T1CCT,Period 1 Day 7,n=3,3: number analyzed (Participants) | 3 | 3
  T1CCT,Period 1 Day 7,n=3,3 | -0.0133 (0.03774) | -0.1250 (0.16975)
  T1CCT,Period 2 Day 7,n=3,3: number analyzed (Participants) | 3 | 3
  T1CCT,Period 2 Day 7,n=3,3 | -0.0343 (0.12948) | -0.0447 (0.11186)

25. Secondary Outcome: Change From Baseline in Chemistry: N-terminal Pro-Brain Natriuretic Peptide
Description: Blood samples were collected to analyze the Chemistry parameter N-terminal pro-Brain Natriuretic Peptide. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline is calculated by subtracting the baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Nanograms per liter
  Period 1 Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1 Day 7,n=5,6 | -279.0 (455.83) | 214.2 (702.54)
  Period 2 Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2 Day 7,n=6,5 | -347.7 (1134.08) | -121.6 (340.70)

26. Secondary Outcome: Change From Baseline in Hematology: Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, White Blood Cell (WBC) Count, Total Neutrophils
Description: Blood samples were collected to analyze the Hematology parameters including Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet count, White Blood Cell (WBC) count, Total Neutrophils. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Giga cells per liter
  Basophils,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Basophils,Period 1, Day 4,n=5,6 | 0.004 (0.0089) | 0.007 (0.0320)
  Basophils,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Basophils,Period 1, Day 7,n=5,6 | 0.000 (0.0100) | 0.010 (0.0358)
  Basophils,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Basophils,Period 2, Day 4,n=5,5 | -0.002 (0.0110) | 0.002 (0.0130)
  Basophils,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Basophils,Period 2, Day 7,n=6,5 | 0.002 (0.0098) | -0.004 (0.0089)
  Eosinophils,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Eosinophils,Period 1, Day 4,n=5,6 | 0.042 (0.0239) | 0.033 (0.0859)
  Eosinophils,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Eosinophils,Period 1, Day 7,n=5,6 | 0.058 (0.0512) | 0.038 (0.0412)
  Eosinophils,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Eosinophils,Period 2, Day 4,n=5,5 | -0.012 (0.0482) | -0.022 (0.0920)
  Eosinophils,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Eosinophils,Period 2, Day 7,n=6,5 | -0.007 (0.0301) | -0.018 (0.1154)
  Lymphocytes,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Lymphocytes,Period 1, Day 4,n=5,6 | 0.128 (0.2876) | -0.110 (0.4315)
  Lymphocytes,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Lymphocytes,Period 1, Day 7,n=5,6 | 0.054 (0.1014) | -0.122 (0.4964)
  Lymphocytes,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Lymphocytes,Period 2, Day 4,n=5,5 | -0.024 (0.1636) | 0.098 (0.3725)
  Lymphocytes,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Lymphocytes,Period 2, Day 7,n=6,5 | 0.025 (0.1512) | 0.126 (0.2508)
  Monocytes,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Monocytes,Period 1, Day 4,n=5,6 | -0.044 (0.0611) | -0.082 (0.1628)
  Monocytes,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Monocytes,Period 1, Day 7,n=5,6 | 0.006 (0.0853) | 0.012 (0.1700)
  Monocytes,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Monocytes,Period 2, Day 4,n=5,5 | -0.064 (0.1236) | -0.014 (0.1150)
  Monocytes,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Monocytes,Period 2, Day 7,n=6,5 | -0.015 (0.1280) | 0.008 (0.1087)
  Platelet count,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Platelet count,Period 1, Day 4,n=5,6 | -1.0 (9.87) | -3.2 (27.26)
  Platelet count,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Platelet count,Period 1, Day 7,n=5,6 | -0.8 (17.46) | -2.7 (25.23)
  Platelet count,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Platelet count,Period 2, Day 4,n=5,5 | -12.8 (9.36) | 1.0 (12.79)
  Platelet count,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Platelet count,Period 2, Day 7,n=6,5 | -6.7 (21.50) | 9.0 (18.40)
  WBC,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  WBC,Period 1, Day 4,n=5,6 | 0.614 (1.2143) | -0.100 (1.3130)
  WBC,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  WBC,Period 1, Day 7,n=5,6 | 0.034 (0.6344) | 0.250 (0.8118)
  WBC,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  WBC,Period 2, Day 4,n=5,5 | 0.156 (0.6105) | 0.252 (1.0176)
  WBC,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  WBC,Period 2, Day 7,n=6,5 | -0.252 (0.6902) | 0.064 (0.3369)
  Total Neutrophils,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Total Neutrophils,Period 1, Day 4,n=5,6 | 0.472 (1.0817) | 0.043 (0.8491)
  Total Neutrophils,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Total Neutrophils,Period 1, Day 7,n=5,6 | -0.064 (0.6789) | 0.345 (0.4476)
  Total Neutrophils,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Total Neutrophils,Period 2, Day 4,n=5,5 | 0.252 (0.6034) | 0.162 (0.8436)
  Total Neutrophils,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Total Neutrophils,Period 2, Day 7,n=6,5 | -0.267 (0.6555) | -0.080 (0.5928)

27. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected to analyze the Hematology parameter Hematocrit. Change from Baseline is presented for this parameter. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Proportion of red blood cells in blood
  Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 4,n=5,6 | -0.0084 (0.01910) | -0.0092 (0.01641)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | -0.0086 (0.02329) | -0.0045 (0.02336)
  Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, Day 4,n=5,5 | 0.0046 (0.00513) | -0.0138 (0.02905)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | -0.0120 (0.01381) | -0.0164 (0.02519)

28. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood samples were collected to analyze Hemoglobin. Change from Baseline is presented for this parameter. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Gram per liter
  Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 4,n=5,6 | -1.0 (6.67) | -4.3 (7.42)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | 0.8 (10.87) | -2.2 (6.55)
  Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, Day 4,n=5,5 | 1.6 (2.41) | -3.8 (7.85)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | -3.5 (4.93) | -3.4 (7.89)

29. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume
Description: Blood samples were collected to analyze Mean Corpuscle Volume. Change from Baseline is presented for this parameter. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Femtoliters
  Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 4,n=5,6 | 0.20 (1.402) | 0.97 (1.218)
  Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Period 1, Day 7,n=5,6 | -0.92 (1.152) | 0.55 (0.946)
  Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, Day 4,n=5,5 | 0.04 (0.493) | 0.08 (0.926)
  Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Period 2, Day 7,n=6,5 | 0.23 (1.003) | -0.50 (1.086)

30. Secondary Outcome: Change From Baseline in Red Blood Cell Count (RBC) and Reticulocytes
Description: Blood samples were collected to analyze the Hematology parameters including RBC and Reticulocytes. Change from Baseline is presented for these parameters. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Trillion cells per liter
  RBC,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  RBC,Period 1, Day 4,n=5,6 | -0.100 (0.1943) | -0.160 (0.2555)
  RBC,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  RBC,Period 1, Day 7,n=5,6 | -0.056 (0.2637) | -0.083 (0.2700)
  RBC,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  RBC,Period 2, Day 4,n=5,5 | 0.014 (0.0937) | -0.146 (0.2708)
  RBC,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  RBC,Period 2, Day 7,n=6,5 | -0.188 (0.2360) | -0.150 (0.2270)
  Reticulocytes,Period 1, Day 4,n=5,6: number analyzed (Participants) | 5 | 6
  Reticulocytes,Period 1, Day 4,n=5,6 | -0.00148 (0.002167) | -0.00388 (0.012096)
  Reticulocytes,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Reticulocytes,Period 1, Day 7,n=5,6 | 0.00049 (0.004412) | 0.00021 (0.010985)
  Reticulocytes,Period 2, Day 4,n=5,5: number analyzed (Participants) | 5 | 5
  Reticulocytes,Period 2, Day 4,n=5,5 | 0.00367 (0.032819) | 0.00051 (0.007178)
  Reticulocytes,Period 2, Day 7,n=6,5: number analyzed (Participants) | 6 | 5
  Reticulocytes,Period 2, Day 7,n=6,5 | 0.00868 (0.019263) | 0.00086 (0.001831)

31. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin Concentration
Description: Blood samples were collected to analyze Mean Corpuscle Hemoglobin concentration . Change from Baseline is presented for this parameter. Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value. NA indicates data was not available. Standard deviation could not be calculated as a single participant was analyzed at the specified time point
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
grams per liter
  Period 1, Day 4,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1, Day 4,n=3,1 | 8.0 (7.94) | -3.0 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1, Day 7,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1, Day 7,n=3,1 | 13.7 (12.22) | -8.0 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 2, Day 4,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2, Day 4,n=1,3 | -1.0 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 2.7 (6.66)
  Period 2, Day 7,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2, Day 7,n=1,3 | -2.0 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 6.0 (8.66)

32. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin
Description: Blood samples were collected to analyze Mean Corpuscle Hemoglobin. Change from Baseline was presented for this parameter. Day -1 was Baseline and change from Baseline was calculated by subtracting the baseline value from specified time point value. NA indicates data was not available. Standard deviation could not be calculated as a single participant was analyzed at the specified time point
Time Frame: Baseline and up to Day 7 in each treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Picograms
  Period 1, Day 4,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1, Day 4,n=3,1 | 0.70 (0.656) | 0.20 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 1, Day 7,n=3,1: number analyzed (Participants) | 3 | 1
  Period 1, Day 7,n=3,1 | 0.70 (1.044) | -0.20 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated.
  Period 2, Day 4,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2, Day 4,n=1,3 | 0.00 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.27 (0.231)
  Period 2, Day 7,n=1,3: number analyzed (Participants) | 1 | 3
  Period 2, Day 7,n=1,3 | 0.40 (NA) — Number of participants analyzed is 1, Standard Deviation could not be calculated. | 0.33 (0.503)

33. Secondary Outcome: Number of Participants With All Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with AE and SAE are reported.
Time Frame: Up to Day 46
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Participants
  Any AE | 5 | 7
  Any SAE | 0 | 1

34. Secondary Outcome: Change From Baseline in Participant Reported Health Status (SF-36) Acute Score
Description: The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (worst) - 100 (best). Day -1 was Baseline and change from Baseline was calculated by subtracting the Baseline value from specified time point value.
Time Frame: Baseline and Day 7 of each treatment period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | GSK2798745 2.4 mg
Number analyzed (Participants) | 11 | 11
Score on a scale
  Physical Functioning, Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Physical Functioning, Period 1, Day 7,n=5,6 | 3.0 (4.00) | 1.2 (0.75)
  Physical Functioning, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Physical Functioning, Period 2, Day 7,n=5,5 | 1.0 (1.22) | -0.4 (2.19)
  Role-Physical, Period 1, Day 7,n=4,6: number analyzed (Participants) | 4 | 6
  Role-Physical, Period 1, Day 7,n=4,6 | -0.5 (3.11) | 3.7 (3.93)
  Role-Physical, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Role-Physical, Period 2, Day 7,n=5,5 | 2.0 (3.67) | 0.4 (2.70)
  Bodily Pain, Period 1, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Bodily Pain, Period 1, Day 7,n=5,5 | -1.0 (1.41) | -1.2 (1.10)
  Bodily Pain, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Bodily Pain, Period 2, Day 7,n=5,5 | -0.2 (1.10) | 0.4 (1.14)
  General Health,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  General Health,Period 1, Day 7,n=5,6 | 1.8 (2.49) | -1.5 (5.79)
  General Health,Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  General Health,Period 2, Day 7,n=5,5 | 0.0 (0.71) | -1.4 (2.97)
  Vitality, Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Vitality, Period 1, Day 7,n=5,6 | 1.2 (1.79) | -1.2 (1.17)
  Vitality, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Vitality, Period 2, Day 7,n=5,5 | -0.4 (1.14) | -0.8 (2.17)
  Social Functioning, Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Social Functioning, Period 1, Day 7,n=5,6 | -0.6 (0.55) | 0.5 (1.22)
  Social Functioning, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Social Functioning, Period 2, Day 7,n=5,5 | 0.6 (0.89) | -0.2 (1.10)
  Role- Emotional, Period 1, Day 7,n=4,6: number analyzed (Participants) | 4 | 6
  Role- Emotional, Period 1, Day 7,n=4,6 | 1.3 (2.50) | 1.0 (1.55)
  Role- Emotional, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Role- Emotional, Period 2, Day 7,n=5,5 | -0.2 (3.19) | 1.2 (4.09)
  Mental Health, Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Mental Health, Period 1, Day 7,n=5,6 | 0.6 (0.55) | 0.3 (0.52)
  Mental Health, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Mental Health, Period 2, Day 7,n=5,5 | 0.2 (1.79) | 1.2 (1.79)
  Physical Health Score,Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Physical Health Score,Period 1, Day 7,n=5,6 | 5.8 (8.23) | 1.7 (3.83)
  Physical Health Score,Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Physical Health Score,Period 2, Day 7,n=5,5 | 2.8 (3.03) | -1.0 (5.61)
  Mental Health Score, Period 1, Day 7,n=5,6: number analyzed (Participants) | 5 | 6
  Mental Health Score, Period 1, Day 7,n=5,6 | 5.2 (6.53) | 0.7 (1.97)
  Mental Health Score, Period 2, Day 7,n=5,5: number analyzed (Participants) | 5 | 5
  Mental Health Score, Period 2, Day 7,n=5,5 | 0.2 (4.09) | 1.4 (3.85)

35. Secondary Outcome: Area Under the Concentration Time Curve (AUC) Time Zero to the Last Time of the Last Quantifiable Concentration (AUC(0-t)), AUC Over the Dosing Interval After First and Last Dose (AUC(0-tau)) and AUCall for GSK2798745
Description: AUC(0-t), AUC(0-tau) and AUCall for GSK2798745 were determined based on intensive Pharmacokinetic (PK) sampling at the following time points: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours on Day 1, pre-dose and at 12 hours post dose on Day 2, pre-dose on Days 3 to 6, Pre-dose, 0.5, 1, 1.5, 2, 3, 5 and 10 hours on Day 7 and at 24 and 48 hours. PK parameter population included all participants in the PK Concentration Population for whom valid and evaluable pharmacokinetic parameters were derived
Time Frame: Day 1 (Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours post-dose), Day 2 (pre-dose, 12 hours post-dose), Days 3 to 6 (pre-dose), Day 7 (Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 10, 24 and 48 hours post-dose)
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per mL
Arm/Group | GSK2798745 2.4 mg
Number analyzed (Participants) | 11
hour*nanogram per mL
  AUC(0-tau), Period 1, Day 1,n=6: number analyzed (Participants) | 6
  AUC(0-tau), Period 1, Day 1,n=6 | 128.3513 (70.4)
  AUC(0-tau), Period 1, Day 7,n=5: number analyzed (Participants) | 5
  AUC(0-tau), Period 1, Day 7,n=5 | 202.2948 (132.1)
  AUC(0-tau), Period 2, Day 1,n=5: number analyzed (Participants) | 5
  AUC(0-tau), Period 2, Day 1,n=5 | 137.7473 (38.4)
  AUC(0-tau), Period 2, Day 7,n=5: number analyzed (Participants) | 5
  AUC(0-tau), Period 2, Day 7,n=5 | 274.0828 (70.9)
  AUCall, Period 1, Day 1,n=6: number analyzed (Participants) | 6
  AUCall, Period 1, Day 1,n=6 | 127.9049 (70.4)
  AUCall Period 1, Day 7,n=5: number analyzed (Participants) | 5
  AUCall Period 1, Day 7,n=5 | 174.7273 (121.5)
  AUCall Period 2, Day 1,n=5: number analyzed (Participants) | 5
  AUCall Period 2, Day 1,n=5 | 137.5038 (38.4)
  AUCall, Period 2, Day 7,n=5: number analyzed (Participants) | 5
  AUCall, Period 2, Day 7,n=5 | 269.0902 (70.5)
  AUC(0-t), Period 1, Day 1,n=6: number analyzed (Participants) | 6
  AUC(0-t), Period 1, Day 1,n=6 | 127.9049 (70.4)
  AUC(0-t) Period 1, Day 7,n=5: number analyzed (Participants) | 5
  AUC(0-t) Period 1, Day 7,n=5 | 174.7273 (121.5)
  AUC(0-t) Period 2, Day 1,n=5: number analyzed (Participants) | 5
  AUC(0-t) Period 2, Day 1,n=5 | 137.5038 (38.4)
  AUC(0-t), Period 2, Day 7,n=5: number analyzed (Participants) | 5
  AUC(0-t), Period 2, Day 7,n=5 | 269.0902 (70.5)

36. Secondary Outcome: Maximum Drug Concentration (Cmax) for GSK2798745
Description: Blood samples for PK analysis were collected at pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours on Day 1, pre-dose and at 12 hours post dose on Day 2, pre-dose on Days 3 to 6, Pre-dose, 0.5, 1, 1.5, 2, 3, 5 and 10 hours on Day 7 and at 24 and 48 hours on Days 8 and 9. Cmax was defined as maximum observed plasma concentration of drug.
Time Frame: as for outcome 35
Population: PK Parameter. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GSK2798745 2.4 mg
Number analyzed (Participants) | 11
Nanograms per milliliter
  Period 1, Day 1,n=6: number analyzed (Participants) | 6
  Period 1, Day 1,n=6 | 10.214 (36.3)
  Period 1, Day 7,n=5: number analyzed (Participants) | 5
  Period 1, Day 7,n=5 | 15.687 (73.6)
  Period 2, Day 1,n=5: number analyzed (Participants) | 5
  Period 2, Day 1,n=5 | 10.017 (48.3)
  Period 2, Day 7,n=5: number analyzed (Participants) | 5
  Period 2, Day 7,n=5 | 15.428 (68.1)

37. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for GSK2798745
Description: Blood samples for PK analysis were collected at pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours on Day 1, pre-dose and at 12 hours post dose on Day 2, pre-dose on Days 3 to 6, Pre-dose, 0.5, 1, 1.5, 2, 3, 5 and 10 hours on Day 7 and at 24 and 48 hours on Days 8 and 9. Tmax was defined as time to maximum observed plasma concentration of drug.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK2798745 2.4 mg
Number analyzed (Participants) | 11
Hour
  Period 1, Day 1,n=6: number analyzed (Participants) | 6
  Period 1, Day 1,n=6 | 3.0 [2 to 3]
  Period 1, Day 7,n=5: number analyzed (Participants) | 5
  Period 1, Day 7,n=5 | 3.0 [1 to 3]
  Period 2, Day 1,n=5: number analyzed (Participants) | 5
  Period 2, Day 1,n=5 | 3.0 [3 to 12]
  Period 2, Day 7,n=5: number analyzed (Participants) | 5
  Period 2, Day 7,n=5 | 2.0 [1 to 3]

38. Secondary Outcome: Elimination Half Life (T½) for GSK2798745
Description: Blood samples for PK analysis were planned to be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8 and 12 hours on Day 1, pre-dose and at 12 hours post dose on Day 2, pre-dose on Days 3 to 6, Pre-dose, 0.5, 1, 1.5, 2, 3, 5 and 10 hours on Day 7 and at 24 and 48 hours on Days 8 and 9. T½ was defined as Elimination half life of drug. Data is not available for t1/2. The analysis was planned but not performed. PK sampling scheme was not adequate enough to reliably estimate the t1/2 of GSK2798745.
Time Frame: as for outcome 35
Population: PK Parameter Population. Data is not available for t1/2. The analysis was planned but not performed. PK sampling scheme was not adequate enough to reliably estimate the t1/2 of GSK2798745.
Arm/Group | GSK2798745 2.4 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the start of study treatment until follow-up (Up to 46 days)
Description: All subject population was used to collect adverse events.
Arm/Group | Placebo | GSK2798745 2.4 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/11
Other Adverse Events (participants affected / at risk) | 5/11 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | GSK2798745 2.4 mg (N=11)
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | GSK2798745 2.4 mg (N=11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02497937/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02497937/SAP_001.pdf